CLINICAL TRIAL: NCT06758804
Title: Evaluation of the Efficacy of Winterized Pistacia Lentiscus Oil in Reducing Purulent Bacterial Overinfection of Pediatric Rhinitis: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy of Winterized Pistacia Lentiscus Oil in Reducing Purulent Bacterial Overinfection of Pediatric Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Experimental Medicine and Clinical Biochemistry, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 116_22.11.2024_BACTORINOL_Siti
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Rhinitis Acute
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Winterized Pistacia Lentiscus Oil Drops (Experimental)
  Interventions: Device: Winterized Pistacia Lentiscus Oil Nasal Drops (Bactorinol®)
- Saline Placebo Drops (Placebo Comparator)
  Interventions: Device: Saline Solution (0.9% NaCl)

INTERVENTIONS:
Device: Winterized Pistacia Lentiscus Oil Nasal Drops (Bactorinol®) — Participants will receive winterized Pistacia lentiscus oil nasal drops (Bactorinol®), administered as 3 drops per nostril, three times daily for six consecutive days.
  Arms: Winterized Pistacia Lentiscus Oil Drops
Device: Saline Solution (0.9% NaCl) — Participants will receive a saline solution (0.9% NaCl) administered as 3 drops per nostril, three times daily for six consecutive days.
  Arms: Saline Placebo Drops

SUMMARY:
This study aims to evaluate the efficacy and safety of a medical device containing winterized Pistacia lentiscus oil in reducing symptoms of purulent bacterial overinfection in pediatric rhinitis and the need for antibiotic therapy. The randomized controlled trial will compare the treatment group receiving nasal drops with a control group using saline solution.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial to assess the therapeutic potential of winterized Pistacia lentiscus oil (WLO) in pediatric patients aged 2 to 10 years with purulent rhinitis. The study will investigate the reduction of rhinitis symptoms, the need for antibiotics, and secondary outcomes including nasal decongestant activity and treatment safety.

Participants will be randomized into two groups: the intervention group will receive 3 drops of WLO per nostril, three times daily for six days, while the control group will use 0.9% saline solution under the same regimen. Clinical evaluations will be conducted by medical staff and parents over six days to record symptom improvement, antibiotic use, and adverse events. The results will contribute to understanding the potential of WLO as a non-antibiotic treatment option for purulent bacterial overinfection in pediatric rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 10 years.
* Clinical symptoms of dense mucosal rhinitis/purulent mucus.
* Onset of symptoms ≤ 5 days before enrollment.

Exclusion Criteria:

* Onset of symptoms > 5 days before enrollment.
* Presence of neurological, malformative, or immunological pathology.
* Suspected or confirmed allergy to the active substance.
* Use of antibiotics within 48 hours prior to enrollment.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Purulent Rhinitis Symptoms | 6 days
  Evaluate the change in symptoms of purulent rhinitis, such as nasal congestion and mucosal discharge, in the experimental group compared to the control group.

SECONDARY OUTCOMES:
Change in Antibiotic Use | 6 days
  Measure the percentage of participants experiencing a change in antibiotic therapy requirements in the experimental group compared to the control group.
Change in nasal obstruction | 6 days
  Change in the nasal obstruction measured via a 10-point Visual Analog Scale.
Incidence of Treatment-Emergent Adverse Events | 6 days
  Record the number and type of treatment-emergent adverse events (TEAEs) related to the use of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi dell'Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arroll B, Kenealy T. Are antibiotics effective for acute purulent rhinitis? Systematic review and meta-analysis of placebo controlled randomised trials. BMJ. 2006 Aug 5;333(7562):279. doi: 10.1136/bmj.38891.681215.AE. Epub 2006 Jul 21. PMID 16861253
- [Background] Orru G, Demontis C, Mameli A, Tuveri E, Coni P, Pichiri G, Coghe F, Rosa A, Rossi P, D'hallewin G. The Selective Interaction of Pistacia lentiscus Oil vs. Human Streptococci, an Old Functional Food Revisited with New Tools. Front Microbiol. 2017 Oct 24;8:2067. doi: 10.3389/fmicb.2017.02067. eCollection 2017. PMID 29114245
- [Background] Di Pierro F, Sagheddu V, Galletti S, Forti M, Elli M, Bertuccioli A, Gaeta S. Antibacterial Activity of a Fractionated Pistacia lentiscus Oil Against Pharyngeal and Ear Pathogens, Alone or in Combination With Antibiotics. Front Microbiol. 2021 Jun 17;12:686942. doi: 10.3389/fmicb.2021.686942. eCollection 2021. PMID 34220777